CLINICAL TRIAL: NCT01343875
Title: Evaluation the Operative Procedure Among Patients That Suffer From Tear of the Distal Tendon of the Biceps
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Shaul Beyth
Other Study IDs: beyth03-HMO-CTIL
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Biceps Tendon Rupture

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- surgery, biceps tear
  Interventions: Procedure: tear of the distal tendon in the biceps muscle

INTERVENTIONS:
Procedure: tear of the distal tendon in the biceps muscle

SUMMARY:
Background: rupture of the distal tendon in biceps muscle is a rare injury. The state of the art treatment is surgical procedure.

Objective: Evaluation of the Surgical procedure among patients that suffered from Methods: The investigators will review files from 2003-2010 of patients that gone through the operation. The investigators will record pre-operation and post-operation process including complications and rehabilitation. The investigators will invite them to the clinic for exams, clinical questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1.see population description

Exclusion Criteria:

1. Unwillingness to come to the clinic visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men and women that went to surgery due to tear of the distal tendon in the biceps muscle.
Sampling Method: Non-Probability Sample